CLINICAL TRIAL: NCT01007539
Title: Efficacy and Safety of CDP-choline in Patients With Methamphetamine Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, MD, PhD, MMS, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KC09MISI0166
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Cytidine Diphosphate Choline; Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDP-choline (Experimental)
  Interventions: Dietary Supplement: CDP-choline
- Placebo (fructose) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo (fructose)

INTERVENTIONS:
Dietary Supplement: CDP-choline — The subjects will be given 1g citicoline twice daily for a total of 8 weeks.
  Arms: CDP-choline
Dietary Supplement: Placebo (fructose) — The Subjects will be given 2 tablets of placebo twice daily for 8 weeks. They will be taking the same quantity as the CDP-choline group.
  Arms: Placebo (fructose)

SUMMARY:
The purpose of the study is to determine if cytidine 5'diphosphocholine (CDP-choline, a naturally occurring chemical in your body) has efficacy in reducing the methamphetamine craving of the subjects with methamphetamine dependence craving and helping them maintain the abstinence. In addition, investigators will measure the brain N-acetyl aspartate (a biologic marker for neuronal viability) level of participants to determine if brain deficits induced by methamphetamine may recover by taking CDP-choline.

ELIGIBILITY:
Inclusion Criteria:

* 19-60 year-old male or female
* Methamphetamine dependence diagnosed by DSM-IV
* Total cumulative dose for methamphetamine during the last two years: over 10 gram (over 200 shots of 0,05 mgram intravenous methamphetamine injection)
* Methamphetamine use in recent 4 weeks
* Subscale score of drug use in ASI: >2

Exclusion Criteria:

* Significant current or past medical, neurological, or psychiatric co-morbidity including cardiovascular, renal, and endocrine disorder, as identified by medical history
* Lifetime axis I psychiatric disorders of bipolar disorder, schizophrenia, identified by SCID-IV
* Socially dysfunctional antisocial personality disorder
* Current alcohol or nicotine dependence identified by SCID-IV
* Taking psychotropic medication in recent two months
* Head trauma history with loss of consciousness or seizure
* Intelligence quotient < 80
* Pregnant subjects. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded. Female subjects who are of child-bearing potential will have to pass a urine pregnancy test before each visit.
* Any contraindication to an MR scan

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Urinary drug screening test | 0-8 week visits

SECONDARY OUTCOMES:
Craving symptoms | 0-8 week visits
Depressive symptoms | 0-8 week visits
Anxiety symptoms | 0-8 week visits
Side effect check | 1-8 week visits
Neuropsychological test battery | 0, 8 week visits
Clinical Global Impression | 0-8 week visits
Alcohol and tobacco use | 0, 4, 8 week visits
Addiction severity index | 0, 8 week visits
Withdrawal symptoms | 0-8 week visits
Magnetic Resonance Scan | 0, 8 week visits
Self-reported drug diary | 0-8 week visits

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul